CLINICAL TRIAL: NCT02196831
Title: Tesamorelin Effects on Liver Fat and Histology in HIV: A Collaborative UO1 Grant
Brief Title: Tesamorelin Effects on Liver Fat and Histology in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1U01AI115711 (NIH); U01AI115711 (NIH)
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Human Immunodeficiency Virus (HIV); Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH)
Keywords: Human immunodeficiency virus (HIV); Nonalcoholic fatty liver disease (NAFLD); Nonalcoholic steatohepatitis (NASH); Growth hormone releasing hormone; tesamorelin
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Non-alcoholic Fatty Liver Disease | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tesamorelin (Experimental): tesamorelin 2mg subcutaneously daily x 12 months double-blind phase. At the end of 12 months, subjects enter open-label tesamorelin treatment phase for 6 months.
  Interventions: Drug: tesamorelin
- Placebo (Placebo Comparator): placebo subcutaneously daily x 12 months double-blind phase. At the end of 12 months, subjects enter open-label tesamorelin treatment phase for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tesamorelin
  Other Names: Egrifta
  Arms: Tesamorelin
Drug: Placebo — inactive substance that looks like tesamorelin
  Arms: Placebo

SUMMARY:
Liver disease is one of the leading co-morbidities of human immunodeficiency virus (HIV) infection, and nonalcoholic fatty liver disease (NAFLD) is present in approximately 30-40% of patients with HIV infection. Nonalcoholic steatohepatitis (NASH) is a more severe form of NAFLD in which increased liver fat is also accompanied by inflammation, cellular damage, and fibrosis.

NAFLD is most prevalent in patients who also have increased visceral adiposity, and our group has previously shown that HIV-infected individuals with increased visceral adiposity generally have decreased growth hormone secretion. Tesamorelin is a growth hormone releasing hormone (GHRH) analogue that increases endogenous growth hormone secretion. Tesamorelin is FDA-approved for the reduction of visceral fat in HIV-infected individuals. In a previous study, treatment with tesamorelin in HIV-infected individuals selected for abdominal adiposity reduced liver fat. The current study is designed to test the effect of tesamorelin on liver fat and steatohepatitis in HIV-infected individuals who have NAFLD. The investigators hypothesize that tesamorelin will reduce liver fat and will also ameliorate the inflammation, fibrosis, and hepatocellular damage seen in conjunction with NASH.

ELIGIBILITY:
Inclusion criteria:

* Men and women 18-70yo
* HIV-infection and treatment with a stable antiretroviral regimen for ≥ 6 months
* Hepatic steatosis as demonstrated by liver fat fraction ≥5% on 1H-MRS
* Hepatitis C antibody negative, or, if Hepatitis C antibody positive, either: a) known clinical disease, successful therapy ≥1 year prior to baseline and undetectable HCV RNA, or b) HCV resolved spontaneously and undetectable HCV RNA. Hepatitis B surface antigen negative at screen visit
* For females ≥50yo, negative mammogram within 1 year of baseline visit
* If use of Vitamin E ≥400 IU daily (in any formulation), stable dose for ≥6 months prior to study.

Exclusion criteria:

* Heavy alcohol use defined as consumption of more than 20g daily for women or more than 30g daily for men for at least 3 consecutive months over the past 5 years
* Use of insulin or thiazoledinediones (TZDs), or HbA1c ≥7%. Individuals with mild diabetes that is well-controlled with diet and/or oral anti-diabetic agents besides TZDs will be included. Use of oral anti-diabetics must have been stable for ≥6 months prior to study entry.
* Known diabetic retinopathy.
* Known cirrhosis, or Child-Pugh score ≥7, stage 4 fibrosis on biopsy, or clinical evidence of cirrhosis or portal hypertension on imaging or exam.
* Chronic corticosteroid use except intermittent use of topical steroid creams and/or prior short-term physiologic corticosteroid use in the ≤ 6 months prior to baseline visit
* Chronic use of methotrexate, amiodarone, or tamoxifen
* Known diagnosis of Alpha-1 antitrypsin deficiency, Wilson's disease, hemochromatosis, or autoimmune hepatitis
* Use of GH or GHRH within the past 1 year
* Change in lipid lowering or anti-hypertensive regimen within 3 months of screening
* HgB < 11.0 g/dL, CD4 < 100 th/mm3, or HIV viral load > 400 copies/mL
* Active malignancy
* For men, history of prostate cancer or evidence of prostate malignancy by PSA > 5 ng/mL
* Severe chronic illness judged by the investigator to present a contraindication to participation
* History of hypopituitarism, head irradiation or any other condition known to affect the GH axis
* Use of physiologic testosterone (men) or estrogen or progesterone (women) unless stable use for a year or more prior to study entry
* Routine MRI exclusion criteria such as the presence of a pacemaker or cerebral aneurysm clip
* Previous weight loss surgery
* For women, positive pregnancy test performed in a CLIA certified laboratory using a test with a sensitivity of at least 25mIU/mL, or breastfeeding.
* Known hypersensitivity to tesamorelin or mannitol
* Unwillingness to abstain from the conception process during the study (i.e., must agree not to participate in an active attempt to become pregnant or impregnate, donate sperm, or participate in in vitro fertilization)
* Unwillingness to use one (for males) or two (for females) reliable methods of contraception while engaging in heterosexual intercourse during the study. Acceptable methods for women include hormonal contraception (estrogen/progesterone or progesterone-only formulations) if stable for a year or more prior to study entry, intrauterine device, or barrier methods (condom, or diaphragm with spermicide). Acceptable methods for males include condom use. This requirement does not apply to women who have been post-menopausal for at least 24 consecutive months or have undergone surgical sterilization, or to men who have undergone surgical sterilization or have documented azoospermia.
* Not willing or able to adhere to dose schedules and required procedures per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — MGH
Locations (2):
- United States (2):
  - National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Stanley TL, Fourman LT, Feldpausch MN, Purdy J, Zheng I, Pan CS, Aepfelbacher J, Buckless C, Tsao A, Kellogg A, Branch K, Lee H, Liu CY, Corey KE, Chung RT, Torriani M, Kleiner DE, Hadigan CM, Grinspoon SK. Effects of tesamorelin on non-alcoholic fatty liver disease in HIV: a randomised, double-blind, multicentre trial. Lancet HIV. 2019 Dec;6(12):e821-e830. doi: 10.1016/S2352-3018(19)30338-8. Epub 2019 Oct 11. PMID 31611038
- [Derived] Fourman LT, Stanley TL, Billingsley JM, Sui SJH, Feldpausch MN, Boutin A, Zheng I, McClure CM, Corey KE, Torriani M, Kleiner DE, Hadigan CM, Chung RT, Grinspoon SK. Delineating tesamorelin response pathways in HIV-associated NAFLD using a targeted proteomic and transcriptomic approach. Sci Rep. 2021 May 18;11(1):10485. doi: 10.1038/s41598-021-89966-y. PMID 34006921
- [Derived] Stanley TL, Fourman LT, Wong LP, Sadreyev R, Billingsley JM, Feldpausch MN, Zheng I, Pan CS, Boutin A, Lee H, Corey KE, Torriani M, Kleiner DE, Chung RT, Hadigan CM, Grinspoon SK. Growth Hormone Releasing Hormone Reduces Circulating Markers of Immune Activation in Parallel with Effects on Hepatic Immune Pathways in Individuals with HIV-infection and Nonalcoholic Fatty Liver Disease. Clin Infect Dis. 2021 Aug 16;73(4):621-630. doi: 10.1093/cid/ciab019. PMID 33852720
- [Derived] Stanley TL, Fourman LT, Zheng I, McClure CM, Feldpausch MN, Torriani M, Corey KE, Chung RT, Lee H, Kleiner DE, Hadigan CM, Grinspoon SK. Relationship of IGF-1 and IGF-Binding Proteins to Disease Severity and Glycemia in Nonalcoholic Fatty Liver Disease. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e520-e533. doi: 10.1210/clinem/dgaa792. PMID 33125080

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject was randomized to tesamorelin but self-discontinued during the baseline visit, prior to receiving any study drug. This individual is included in baseline characteristics but is not counted as starting tesamorelin (hence the discrepancy between 61 total enrolled and the 30 in tesamorelin and 30 in placebo group shown in participant flow).
Groups:
- Tesamorelin: tesamorelin 2mg subcutaneously daily x 12 months double-blind phase. At the end of 12 months, subjects enter open-label tesamorelin treatment phase for 6 months.
  tesamorelin
Period: Overall Study
Arm/Group | Tesamorelin | Placebo
Started | 30 | 30
Received Follow-up Imaging | 26 | 28
Completed | 21 | 26
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Population: All randomized patients. One patient in the tesamorelin group discontinued before receiving study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesamorelin | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 54 (7) | 53 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White (all ethnicities) | 21 | 19 | 40
  Race: Black (all ethnicities) | 8 | 10 | 18
  Race: Other (all ethnicities) | 2 | 1 | 3
Hepatic Fibrosis Stage [Count of Participants; unit: Participants] — Fibrosis Stage is determined through standardized histological grading by pathologists; this measure is used routinely in evaluation of patients with liver disease. Stage 1 is the mildest fibrosis, and Stage 4 represents cirrhosis. Those unfamiliar can find a review of this staging system in Kleiner DE and Brunt EM, Nonalcoholic Fatty Liver Disease: Pathologic Patterns and Biopsy Evaluation in Clinical Research, 2012, Semin Liver Dis, 32:003-013.
  Participants
    Stage 0 (No Fibrosis) | 15 | 18 | 33
    Stage 1 Fibrosis | 4 | 5 | 9
    Stage 2 Fibrosis | 6 | 4 | 10
    Stage 3 Fibrosis | 4 | 2 | 6
    Data Not Available | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Fat as Measured by 1-H Magnetic Resonance Spectroscopy
Description: change (value at 12 months minus value at baseline). Hepatic fat fraction is a standardized measure used to describe the percent fat in the liver. As it is determined by spectroscopy, it is quantified by the area under the lipid peak, standardized to the total area under the (lipid peak + water peak). Using 1-H Magnetic resonance spectroscopy to quantify liver fat in this manner was first described by Longo R et al., Invest Radiol, 1993, 28(4):297-302.
Time Frame: change between baseline and 12 months
Population: These are participants who had magnetic resonance spectroscopy for hepatic fat fraction at 0 and 12 months. This is different from the primary analysis population reported in the manuscript.
Measure: Mean (Standard Deviation); unit: percent (hepatic fat fraction)
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 20 | 25
percent (hepatic fat fraction) | -4.7 (6.6) | 0.0 (4.1)

2. Secondary Outcome: Change in Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score
Description: change (value at 12 months minus value at baseline). The nonalcoholic fatty liver disease (NAFLD) activity score is a standardized histological quantification of NAFLD severity designed and validated by the Nonalcoholic Steatohepatitis Clinical Research Network (Kleiner DE et al., Hepatology, 2005, 41(6):1313-1321). The score is the sum of three semi-quantitative histological grades:
  1. steatosis, graded from 0 [<5% liver fat] to grade 3 [>66% liver fat]
  2. lobular inflammation, graded from 0 [no foci of inflammation] to 3 [>4 foci per 200x field]
  3. hepatocellular ballooning, graded from 0 [no ballooning] to 2 [many cells/prominent ballooning] The "total" NAFLD activity score, a sum of the three components below, ranges from 0 to 8, with a higher score generally representing greater severity of NAFLD/nonalcoholic steatohepatitis.
Time Frame: change between baseline and 12 months
Population: all participants with available biopsy data from both baseline and 12 month visits
Measure: Mean (Standard Deviation); unit: score on a scale, NAFLD activity score
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 19 | 24
score on a scale, NAFLD activity score | -0.16 (1.34) | 0.13 (1.03)

3. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: change (value at 12 months minus value at baseline)
Time Frame: change from baseline to 12 months
Population: all participants with available data at both baseline and 12 month visits
Measure: Mean (Standard Deviation); unit: units/liter (U/L)
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 21 | 24
units/liter (U/L) | -2 (11) | 5 (15)

4. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: change (value at 12 months minus value at baseline)
Time Frame: change from baseline to 12 months
Population: all participants with available data at both baseline and 12 month visits
Measure: Mean (Standard Deviation); unit: units/liter (U/L)
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 20 | 24
units/liter (U/L) | -2 (11) | -2 (4)

ADVERSE EVENTS:
Time Frame: Adverse events reported herein are from the double-blind (tesamorelin vs. placebo) phase of the study which was 12 months in length as well as the subsequent open-label phase 6 months in length.
Description: The primary analysis is from baseline to 12 months, during the "double-blind" phase. Adverse events from this phase are reported under the "Tesamorelin (Double-blind phase)" and "Placebo (Double-blind phase)" descriptors. 43 participants subsequently entered a 6 month open label phase during which all received tesamorelin. Data from this phase are not included in analysis, but Adverse Event data from the Open Label phase are included under the descriptor, "Open Label Tesamorelin Arm."
Groups:
- Tesamorelin (Double-blind Phase): tesamorelin 2mg subcutaneously daily x 12 months double-blind phase. At the end of 12 months, subjects enter open-label tesamorelin treatment phase for 6 months.
  tesamorelin
- Placebo (Double-blind Phase): placebo subcutaneously daily x 12 months double-blind phase. At the end of 12 months, subjects enter open-label tesamorelin treatment phase for 6 months.
  Placebo: inactive substance that looks like tesamorelin
- Open Label Tesamorelin Arm: following the 12 month double-blind period, all subjects received open-label tesamorelin 2mg daily subcutaneously for 6 months.
Arm/Group | Tesamorelin (Double-blind Phase) | Placebo (Double-blind Phase) | Open Label Tesamorelin Arm
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 1/43
Serious Adverse Events (participants affected / at risk) | 4/31 | 2/30 | 3/43
Other Adverse Events (participants affected / at risk) | 29/31 | 29/30 | 35/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tesamorelin (Double-blind Phase) (N=31) | Placebo (Double-blind Phase) (N=30) | Open Label Tesamorelin Arm (N=43)
Hemiplegia transient (Nervous system disorders) | 1 | 0 | 0
Anxiety Depression (Psychiatric disorders) | 0 | 0 | 1
Hepatic Hematoma (Hepatobiliary disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 — influenza requiring hospitalization
Drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Active suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Death sudden (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tesamorelin (Double-blind Phase) (N=31) | Placebo (Double-blind Phase) (N=30) | Open Label Tesamorelin Arm (N=43)
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 7 | 5 | 4
Alkaline phosphatase increased (Investigations) | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1
Fasting blood glucose increased (Investigations) | 12 | 11 | 14
Fatigue (General disorders) | 2 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0
Hyper LDL cholesterolemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 3 | 2
Injection site bruising (General disorders) | 11 | 11 | 1
Injection site induration (General disorders) | 3 | 0 | 1
Injection site itching (General disorders) | 4 | 1 | 0
Injection site pain (General disorders) | 2 | 0 | 1
Injection site redness (General disorders) | 4 | 0 | 0
Injection site stinging (General disorders) | 4 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Nonspecific abnormal findings on radiological and other examinations (Investigations) | 1 | 2 | 0
Pain post biopsy (Injury, poisoning and procedural complications) | 3 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 3 | 0
Tooth Infection (Infections and infestations) | 2 | 1 | 1
URTI (upper respiratory tract infection) (Infections and infestations) | 5 | 5 | 3
Viral infection (Infections and infestations) | 1 | 2 | 1
Paresthesia (Nervous system disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02196831/Prot_SAP_000.pdf